CLINICAL TRIAL: NCT02749344
Title: Natural Cycle/Progesterone Fortified Protocol for Endometrial Preparation for Frozen/Thawed Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Amir Weiss, Dr., HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0074-15-EMC
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Infertility
Keywords: Frozen Embryo Transfer, Progesterone, Endometrium
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FET after endometrial preparation (Experimental): Natural cycle/progesterone fortified endometrial preparation before embryo transfer
  Interventions: Other: FET after endometrial preparation

INTERVENTIONS:
Other: FET after endometrial preparation — Patients included in the protocol will begin progesterone supplementation 48 hours before scheduled embryo transfer once it has been established that the endometrium is at least 7 mm and there is a leading follicle.

SUMMARY:
This is a pilot study of a novel protocol for preparation of the endometrium for frozen/thawed embryo transfer whereby estrogen is not administered during the proliferative phase and progesterone is administered through vaginal suppositories in accordance with endometrial thickness only, disregarding the day of ovulation. Progesterone supplementation commences once the endometrium is at least 7 mm, a follicle is demonstrated on TVS, and ovulation has not yet taken place. The day of ET is scheduled according to the unit's working days and progesterone suppositories are commenced 48 hours before the scheduled embryo transfer.

DETAILED DESCRIPTION:
Natural cycle/progesterone fortified protocol for endometrial preparation for frozen/thawed embryo transfer Study type: Descriptive pilot study of a novel protocol for endometrial preparation for frozen/thawed embryo transfer Introduction: In the process of in-vitro fertilization (IVF) cycles embryos are frequently cryopreserved for future attempts at conception. In order for these embryos to take root in the uterus, the endometrial lining must be made "receptive" to embryo implantation.

During the natural reproductive cycle, this process takes place in two stages. During the endometrium's proliferative phase, which takes place during the first 14 days of a 28 day cycle, estradiol is produced by the growing follicle whereby the thin endometrium remaining after the menstrual cycle proliferates to a width of between 7 to 14 mm on average, attains a triphasic appearance on ultrasound and acquires receptors for progesterone. After ovulation, the ovarian follicle transforms to a corpus luteum which produces progesterone. At this stage, exposure to progesterone transforms the endometrium to one which is receptive to embryo implantation. There is a minimum level of progesterone and a minimum time of exposure which is necessary to transform the endometrium to a receptive one while prolonged progesterone exposure renders the endometrium hostile to implantation. The boundaries of this time zone are referred to as the window of implantation. The length of time of this window is unknown.

There are two strategies for returning frozen/thawed embryos to the uterus in women with regular menstrual cycles.

1. The natural cycle: In our facility embryos are cryopreserved 48-72 hours after fertilization. In the natural cycle protocol women are monitored for estradiol, progesterone and LH levels in the blood and endometrial thickness and follicle development. The thawed embryos are transferred to the uterus 48-72 hours after presumed ovulation and the rise of progesterone
2. Hormone replacement protocol: The patient is given beta estradiol 2mg three times a day (Estrofem - Novo Nordisk) from the first day of the menstrual cycle. This prevents indigenous follicle development on the one hand, but is sufficient to prepare the endometrium. When the endometrium is at least 7 mm thick vaginal suppositories of progesterone are administered 100 mg tid (Endometrin - Lapidot) for 48 hours after which the embryos are transferred. If the endometrium fails to reach 7 mm, additional estrogen is added. Since there is no corpus luteum in this protocol, estradiol and progesterone supplementation must be given until the placenta produces these hormones in sufficient quantities. We maintain hormonal support until 11.6 weeks of gestation in cycles where pregnancy is attained.

The advantage of the natural cycle is that there is no need to take hormones. Nevertheless, it should be noted that even though progesterone supplementation is not necessary for the natural cycle protocol, many IVF units add progesterone support after embryo transfer. A recent study demonstrated that adding progesterone to the natural cycle increased the live birth rate (Bjuresten et al. 2011). Patients were monitored from day 10 to 14 for follicular development after which daily home urinary kits were provided to detect the LH surge. Three days after detection of the LH surge thawed embryos were transferred and patients in the study group commenced taking vaginal progesterone.

The disadvantages of the natural cycle is that the IVF unit must be prepared to perform an embryo transfer on every day of the week including days on which the unit is closed, in accordance with the day of ovulation. Delaying embryo transfer to the unit's work schedule may cause the embryo transfer to take place outside of the endometrium's window of implantation.

In the hormone replacement protocol the physician determines the day the patient begins progesterone supplementation, and therefore the day of embryo transfer can be scheduled according to the units work load. Furthermore there is no need for blood tests during patient monitoring. Ultrasound monitoring can usually be limited to two or three visits. The hormone replacement protocol is the protocol of choice in our unit.

Rationale:

Ovulation is not essential for embryo implantation in the endometrial lining as demonstrated in the hormone replacement protocol. In the proposed protocol the developing follicle stimulates endometrial growth and progesterone is commenced once endometrial growth reaches at least 7 mm and the dominant follicle has been established, regardless of when ovulation occurs. Embryo transfer is performed 48 hours after beginning progesterone. By dissociating the protocol from the day of ovulation greater leeway is achieved in choosing the day of embryo transfer.

Objectives:

This is a pilot study of a novel protocol for preparation of the endometrium for frozen/thawed embryo transfer whereby estrogen is not administered during the proliferative phase and progesterone is administered through vaginal suppositories in accordance with endometrial thickness only, disregarding the day of ovulation. The primary outcome is the biochemical pregnancy rate. Secondary outcomes include the clinical pregnancy rate and ongoing pregnancy rate.

Intervention: We propose a protocol for endometrial preparation for frozen/thawed embryo transfer which combines the advantages of both protocols. Patients do not receive estradiol and therefore ovarian follicle production is not suppressed. Progesterone supplementation commences once the endometrium is at least 7 mm, a follicle is demonstrated on TVS, and ovulation has not yet taken place. The day of ET is scheduled according to the unit's working days and progesterone suppositories are commenced 48 hours before the scheduled embryo transfer. In order to ensure synchronization between the endometrium and the embryos, embryo transfer of 48 hour embryos will be transferred 48 hours after progesterone therapy. This is not different from our current practice.

Like the natural cycle protocol, we allow ovulation to take place but we are not dependent on the day of ovulation to dictate to us the day of embryo transfer, as long as we begin progesterone supplementation before or at the same time as the natural rise of progesterone which accompanies ovulation. The progesterone supplementation dose is identical to the standard protocol so that even if ovulation is suppressed the luteal support is adequate.

In this protocol there is no need for daily blood and ultrasound studies. For most patients, one visit around day 10-13 will probably suffice to schedule the embryo transfer. Progesterone supplementation can be less intensive and estrogen supplementation unnecessary.

Recruitment:

Recruitment for the study will be done by the investigators who are all senior ob/gyn specialists at the IVF unit. Patients to be recruited are those women who have cryopreserved embryos in our unit and who request a frozen thawed embryo replacement cycle. No recruitment outside of the unit will take place, no transfer of frozen embryos from other units will be included and therefore no advertising is necessary.

Inclusion criteria:

1. Women younger than 39 at the time of cryopreservation
2. Regular menstrual cycles of at least 26 days and at most 32 days.
3. Women with no more than 3 failed prior embryo transfers
4. Patients with embryos cryopreserved 48 hours after ovum pick up Exclusion and withdrawal criteria

1. Women with known uterine malformations or significant myomas 2. Women with elevated Progesterone of at least 1.5 ng/mL for the duration of more than 72 hours before embryo transfer can be performed 3. Women suspected of having endometrial pathology based on previous treatment cycles i.e. "thin endometrium", polyps, adhesions 4. Women whose embryos did not survive the thawing process, i.e. no embryos available for transfer after thawing 5. Women without follicular development

Protocol:

A blood sample for estradiol, progesterone and LH will be taken on days 10 - 14 of a 28 day cycle as well as a TVS study of the endometrial thickness and ovarian follicles. The day of the first visit can be adjusted according to the length of the cycle.

Based on these tests the physician will determine if there is active follicle formation prior to ovulation. Evidence of active follicle formation includes a clear follicle of at least 12 mm and estradiol of at least 80 pg/ml. If the endometrium is at least 7 mm, ET will be scheduled. If the endometrium is less than 7 mm the patient will be invited for a second visit 1-3 days later.

Should there be evidence of ovulation having already taken place, such as a progesterone level over 1.5 ng/ml and sonographic evidence of a corpus luteum, then the cycle will be cancelled.

If there is no evidence of follicular activity at the first visit after menstruation; i.e. estradiol under 80 pg/ml and no follicle demonstrated on ultrasound, the patient will be withdrawn from the study.

Progesterone suppositories (Endometrin), 100 mg 3 times a day will commence 48 hours before scheduled embryo transfer until the day of the pregnancy test 14 days later. All embryo transfers will be done under abdominal ultrasound guidance. At the time of embryo we will record the size of the leading follicle and whether it has attributes of a corpus luteum.

Once pregnancy is confirmed progesterone support will be continued until 11.6 weeks three times a day. Blood samples and sonographic studies will be done as needed until embryo transfer. HCG, progesterone and estradiol will be measured 14 days after embryo transfer and 16-17 days after should a pregnancy be detected. An ultrasound will be performed at 5-6 weeks to confirm the presence of a gestational sac and at 6-7 weeks to confirm a heartbeat. Data will be collected until pregnancy termination or delivery.

Sample size:

The biochemical pregnancy rate for FET in our unit for patients of this age group is 24%.

A sample size of 40 patients will provide 13% accuracy for pregnancy rate. Recruitment will end after 40 patients have completed the protocol up to the stage of embryo transfer. Up to 75 women will be recruited in order to assure that 40 patients complete the protocol. The primary endpoint is the biochemical pregnancy rate. Secondary endpoints include implantation rate and clinical pregnancy rate. For the purposes of comparison a cohort of patients not in the study undergoing the traditional hormone replacement preparation will be analyzed.

All patient data will be kept confidential by all researchers. Patient research files will be kept in a locked closet in the IVF unit. Patients names and ID numbers will be replaced by patient codes in the database before submitting for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Women younger than 39 at the time of cryopreservation
2. Regular menstrual cycles of at least 26 days and at most 32 days.
3. Women with no more than 3 failed prior embryo transfers
4. Patients with embryos cryopreserved 48 hours after ovum pick up

Exclusion Criteria:

1. Women with known uterine malformations or significant myomas
2. Women with elevated Progesterone of at least 1.5 ng/mL for the duration of more than 72 hours before embryo transfer can be performed
3. Women suspected of having endometrial pathology based on previous treatment cycles i.e. "thin endometrium", polyps, adhesions
4. Women whose embryos did not survive the thawing process, i.e. no embryos available for transfer after thawing
5. Women without follicular development

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Biochemical Pregnancy | 14 days after embryo transfer
  Positive betaHCG blood test

SECONDARY OUTCOMES:
Clinical Pregnancy | 3-4 weeks after embryo transfer
  Ultrasound detection of intrauterine gestational sac
Ongoing Pregnancy | 5 weeks after embryo transfer
  Ultrasound detection of fetal pole and heart rate of at least 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided